CLINICAL TRIAL: NCT03966131
Title: Experimental Study of Tongue/Palate Interactions Using Upper coMplete dEnture
Brief Title: TOngue/Palate Interactions Study
Acronym: EEXPLORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL18_0103
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Toothless
Keywords: Speech; swallowing; sensors; complete denture
MeSH Terms: conditions — Speech

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with complete denture for the first time (Experimental): Arm that allows to follow the adaptation of this population to the new complete denture during the tasks of speech production and swallowing.
  Interventions: Device: Tongue pressure recordings with the PRESLA prothesis for the Arm1 (patients wearing the complete denture for the first time)
- patients with complete denture used to their complete denture. (Experimental): Arm that allows a descriptive cross-sectional study of tongue pressure measurements during the tasks of speech production and swallowing
  Interventions: Device: Tongue pressure recordings with the PRESLA prothesis for the Arm2 (patients used to wear the complete denture)

INTERVENTIONS:
Device: Tongue pressure recordings with the PRESLA prothesis for the Arm1 (patients wearing the complete denture for the first time) — Tongue pressure recordings during speech production, wet and dry swallowing tasks planned in 3 sessions, when the complete denture is worn for the first time, after 3 weeks, then after 3 months in order to characterise the adaptation to this new prosthesis.
  Arms: patients with complete denture for the first time
Device: Tongue pressure recordings with the PRESLA prothesis for the Arm2 (patients used to wear the complete denture) — These measures provide to establish a spatial and temporal mapping of contacts applied by the tongue and lips to the prosthesis during speech production in patients used to their prosthesis. They also provide to establish a spatial and temporal mapping of contacts applied by the tongue and lips to the prosthesis during swallowing) in these patients. The measurement is made at once when the new denture which replaces the old one is placed in the mouth.
  Arms: patients with complete denture used to their complete denture.

SUMMARY:
The project aims to assess the effect of a complete denture of new denture wearers on speech production using sensors placed inside a duplicate of the prosthesis according to the technique described in the PRESLA system. Secondly, it aims to assess the effect of a complete denture on swallowing for these new denture wearers. Thirdly it aims to describe a precise mapping of the mechanical pressures exerted by the tongue on the palate of complete denture user, been used in wearing denture, during speaking and swallowing. The experiments will take place in the department of treatments and dental consultations of the Hospices Civils de Lyon (Faculty of Odontology, Lyon, France).

DETAILED DESCRIPTION:
The evaluation of speech production is based on the characteristics of the pressure signal (time and frequency) and the acoustic signal after synchronization during time using duplicate with up to 8 sensors.

To reach the first objective, the investigators will focus on the patients who wear new complete denture during the first session of recording. They will first analyze the characteristics of the acoustic and pressure signals of the production of consonants. They shall select from 8 sensors, 3 sensors for the inferential analysis: a previous sensor in the alveolar zone, a median sensor in the palatal zone and a posterior sensor in the palatal area (on the border of the beginning of the soft palate). These 3 sensors will be selected on the basis of the amplitude of the variations of pressure during the task. This sensor's triplet will be specific to every patient. The investigators shall thus have after 3 sensors called: previous, median, posterior. They shall do, for every sensor's measurements and for the acoustic measures, an inferential statistical analysis based on one model shelf spaces generalized in mixed effects, in which the variable to be explained will be one of moderate variables, the fixed effects will be the session (just after wearing the prosthesis for the first time, 3 weeks later, 3 months later), the consonant, the index of the sensor (1 - 3, from the front to the back) and the index of the repetition (from 1 to 15), and where the random effect will be the patient.

ELIGIBILITY:
Inclusion Criteria:

* Bimaxillary edentulous patients of both genders, over 18 years of age, requiring prosthesis (Cohort 1).
* Bimaxillary edentulous patients of both genders, over 18 years of age, with prosthesis made since at least one year (Cohort 2).
* Patients Affiliated with the French Social Security Insurance

Exclusion Criteria:

* Patients with speech or neurological disorders, or uncorrected or psychiatric sensory disorders
* Patients without French as native language
* Pregnant women
* Patients deprived of liberty or provided with legal protection
* Patients unable to support study constraints as determined by investigator
* Patients who have expressed their refusal to participate with the investigator
* Allergy to methacrylic resin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Pressure signal (time and amplitude) at week 3 and month 3, during speech production for new denture wearers using duplicate with up to 8 sensors | Day 0 (Baseline), Week 3 and Month 3
  The evaluation of speech production is based on the characteristics of the pressure and acoustic signals after synchronization during time, using duplicate with up to 8 sensors.
Change from Baseline Pressure signal Acoustic signal (time and frequence) at week 3 and month 3, during speech production for new denture wearers using duplicate with up to 8 sensors | Day 0 (Baseline), Week 3 and Month 3
  The evaluation of speech production is based on the characteristics of the pressure and acoustic signals after synchronization during time, using duplicate with up to 8 sensors.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Consultations et de Traitements Dentaires des Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No